CLINICAL TRIAL: NCT06159751
Title: PROGNOSTIC ROLE OF SERUM ALBUMIN LEVEL IN RADIOLOGICAL PROGRESSION OF GONARTHROSIS: IS IT A BIOMARKER IN ITSELF? A BIOMARKER ASSOCIATED WITH SYSTEMIC INFLAMMATION?
Status: Completed | Type: Observational
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Elzem Bolkan Günaydın, MD, Ufuk University
Other Study IDs: 12024861-02
Record Dates: First submitted 2023-11-28; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Gonarthrosis; Serum Albumin Low
MeSH Terms: conditions — Osteoarthritis, Knee; Hypoalbuminemia | interventions — Serum Albumin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: serum albumin level — serum albumin level in gonarthrosis

SUMMARY:
The aim of our study is to evaluate the prognostic roles of serum albumin level and systemic inflammation-related indices, including and not including serum albumin level, in the radiological progression of gonarthrosis. In this retrospective study, between 10.01.2017 and 10.01.2022, the data of the patients between the ages of 50-80, who applied to Ufuk University Physical Medicine and Rehabilitation clinic with the complaint of knee pain and met the clinical criteria of the American Rheumatology Association for gonarthrosis (knee osteoarthritis) (knee pain on many days of the previous month, crepitation with active joint movement, morning stiffness lasting ≤ 30 minutes, age ≥38 years, bone enlargement of the knee on examination),and whose knee radiography and blood tests were evaluated at admission were scanned.

ELIGIBILITY:
Inclusion Criteria:

* In this retrospective study, between 10.01.2017 and 10.01.2022, the data of the patients between the ages of 50-80, who applied to Ufuk University Physical Medicine and Rehabilitation clinic with the complaint of knee pain and met the clinical criteria of the American Rheumatology Association for gonarthrosis (knee osteoarthritis) (knee pain on many days of the previous month, crepitation with active joint movement, morning stiffness lasting ≤ 30 minutes, age ≥38 years, bone enlargement of the knee on examination),and whose knee radiography and blood tests were evaluated at admission were scanned. In order to compare the parameters to be included in the study, the data and blood tests of patients between the ages of 50-80 who applied to Ufuk University Physical Medicine and Rehabilitation clinic between 10.01.2017 and 10.01.2022 for reasons other than knee pain were scanned.

Exclusion Criteria:

* In the patient and control groups, patients who were younger than 50 years of age, older than 80 years of age, had acute or chronic infection, malignancy, rheumatic disease or systemic diseases that could change the blood test parameters to be evaluated, and patients who were missing one or more of the blood test parameters planned to be evaluated among the data obtained were excluded from the study. In addition, in the patient group, patients who had neurogenic or internal organ problems that could cause pain referred to the knees, who were not required to have a knee X-ray when applying to the outpatient clinic, and who had a history of trauma to the knee area, invasive procedure or surgical intervention within the 6 months before admission to the outpatient clinic, were excluded from the study. In the control group, patients who complained of knee pain in addition to their complaints at admission were excluded from the study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: - In this retrospective study, between 10.01.2017 and 10.01.2022, the data of the patients between the ages of 50-80, who applied to Ufuk University Physical Medicine and Rehabilitation clinic with the complaint of knee pain and met the clinical criteria of the American Rheumatology Association for gonarthrosis and whose knee radiography and blood tests were evaluated at admission were scanned. In order to compare the parameters to be included in the study, the data and blood tests of patients between the ages of 50-80 who applied to Ufuk University Physical Medicine and Rehabilitation clinic between 10.01.2017 and 10.01.2022 for reasons other than knee pain were scanned.
Sampling Method: Probability Sample
Enrollment: 375 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
serum albumin level | 1 month
  serum albumin level
The Aggregate Index of Systemic Inflammation (AISI) | 1 month
  Neutrophil countxPlatelet countxMonocyte count/ Lymphocyte count
Systemic Inflammatory Response Index (SIRI) | 1 month
  Neutrophil countxMonocyte count/ Lymphocyte count
Systemic Immune Inflammation Index (SII) | 1 month
  Platelet countxNeutrophil count/Lymphocyte count
Prognostic Nutrisyonel Index (PNI) | 1 month
  Serum albumin concentration (g/l) + (5xlymphocyte count (thousand/microlitre)
Modified Systemic Inflammation Score (mSIS) | 1 month
  Serum albumin concentration <40g/l ve LMR<3.4: score 2 Serum albumin concentration ≥40 g/l veya LMR≥3.4: score 1 Serum albumin concentration ≥40 g/l ve LMR≥3.4: score 0

CONTACTS AND LOCATIONS:
Locations (1):
- Ufuk University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No